CLINICAL TRIAL: NCT04243226
Title: Develop and Rehabilitation Effects of the Safety Aerobic Exercise Prescription on Cognition, Depression and Quality of Life in Traumatic Brain Injury Patients- Taking the Cerebral Blood Circulation As a Mediator
Brief Title: Effects of Aerobic Exercise on Cognition,cerebral Brain Flow and Mental Health Among Traumatic Brain Injury Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hui-Hsun Chiang, Associate Professor, RN, PhD, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 30988
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cardiology; Psychiatry
Keywords: physical health care; Activity of Daily Living,ADL

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: 1. Traumatic brain injury patients with GCS 8-13 and GCS 14-15
  2. Discharged within 3 months
  3. Can communicate and conversation with Mandarin Chinese or Taiwanese
  4. Agree to join the research
  5. Can walk and communicate individually and live in big Taipei area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- this study is to develop exercise prescription of TBI patients (Experimental): The aim of this study is to develop exercise prescription of TBI patients and then to evaluate the effectiveness of programmed aerobic exercise to improve psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life. This will be a randomized-controlled clinical trial, by using a mixed method to explore the feasibility and validity of such a safety exercise prescription. In the next stage, a randomized clinical control trial will be applied in TBI patients to evaluate the effectiveness of programmed aerobic exercise to promote psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life.
  Interventions: Device: telehealth-based aerobic walking exercise
- No exercise prescription in TBI patients (No Intervention): Routine Care of TBI Patients

INTERVENTIONS:
Device: telehealth-based aerobic walking exercise — The aim of this study is to develop exercise prescription of TBI patients and then to evaluate the effectiveness of programmed aerobic exercise to improve psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life.
  Other Names: aerobic exercise; walking exercise; theoretical-based aerobic exercise; walking
  Arms: this study is to develop exercise prescription of TBI patients

SUMMARY:
The aim of this study is to develop exercise prescription of TBI patients and then to evaluate the effectiveness of programmed aerobic walking exercise to improve cognitive performance, depression relief, motivation, symptom, resilience and quality of life with improvement of CBF. This will be a randomized controlled clinical trial, using a mixed method to explore the feasibility and validity of such a safety exercise prescription. Then, a randomized clinical control trial will be applied in TBI patients to evaluate the effectiveness of programmed aerobic exercise to promote psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) brings out the major cause of accidental disability. Aerobic exercise can increase the influx of blood circulation improving cognitive performance, such as walking and cycling. Yet the effective exercise prescription improves cerebral blood flow (CBF) on promoting psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life. PI conducted a retrospective study in TBI patients and results indicated that 93% of patients discharged among 5000 TBI patients in the past decade. However, about 70% TBI outpatients have squeals left by TBI, which not only affect physical activity, cognition, but also cause mental health problems such as depression and also family care burden and huge medical burdens. The preliminary data showed the significant effects of promoting cerebral blood flow (CBF) through aerobic exercise. This study intends to explore the effectiveness of aerobic exercise prescription among patients with TBI on their physical and mental health based on PI's experiences of walking exercise intervention research and their publications.

The aim of this study is to develop exercise prescription of TBI patients and then to evaluate the effectiveness of programmed aerobic exercise to improve psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life with improvement of CBF. This will be a comprehensive randomized controlled clinical trial using a mixed method to explore the feasibility of such a safety exercise prescription. Then, a randomized clinical control trial will be applied in TBI patients to evaluate the effectiveness of programmed aerobic exercise to promote psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life.

First, a concurrent parallel design combining qualitative and quantitative mixed methods approach will be conducted to explore the accuracy and appropriateness of the prescription and predictability of the mental health and user's experiences. We plan to recruit 30 TBI patients who will be intervened with moderate to high intensity aerobic exercise. We will collect informations regarding CBF and cardiac force index (CFI) during the progress of aerobic exercise. Moreover, we will evaluate the psysical-psycho-social health such as cognitive status, 6 minutes walk test, depression relief, motivation, symptom, resilience and quality of life. We will examine the sensitivity, specificity and accuracy of the CFI and CBF monitor system, and to explore the experience of adopting aerobic exercise prescription among TBI patients. Depending on the results of the first two years, the safety aerobic exercise prescription with CFI and CBF monitor system will be modified and piloted in the next stage. We plan to recruit at least 120 patients and randomized them into an intervention group (N=60) that received the aerobic exercise prescription and a control group (N=60) that received usual care. Outcome variables will be followed at the pretest, the first, second, third and sixth month after the exercise prescription has been implemented. Intention-to-treat and multiple linear models will be used to analyze the results. We hope to develop the safety aerobic exercise prescription with empirical evidence of promoting mental health for patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with mild traumatic brain injury at the emergency department
2. GCS score of 14-15 at the emergency department or patients with moderate brain injury (GCS score of 8-13
3. Brain injury Patients more than three months after discharge
4. Can communicate in Chinese and Taiwanese
5. Patients who have good audio-visual ability to complete tests and data filling
6. Patients are willing to sign a consent form to participate in the research.
7. Each subject was able to walk on their own, communicate freely and live in Taipei or Greater Taipei.

Exclusion Criteria:

1. Exclude those with severe impairment of cognition, emotions and executive function caused by prefrontal lobe injury
2. Exclude patients with brain injury due to head puncture.
3. Regularly perform moderate-intensity aerobic exercise.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
cerebral blood flow (CBF)-(T1) | T1_Baseline
  Hemoencephalography (HEG) will be measure by Bioland, the unit is ratio A/B and the brain SPECT
cerebral blood flow (CBF)-(T2) | T2_1 month later
  Hemoencephalography (HEG) will be measure by Bioland, the unit is ratio A/Band
cerebral blood flow (CBF)-(T3) | T3_2 months later
  Hemoencephalography (HEG) will be measure by Bioland, the unit is ratio A/B
cerebral blood flow (CBF)-(T4) | T4_3 months later
  Hemoencephalography (HEG) will be measure by Bioland, the unit is ratio A/B
cerebral blood flow (CBF)-(T5) | T5_6 months later
  Hemoencephalography (HEG) will be measure by Bioland, the unit is ratio A/B and the brain SPECT
cerebral blood flow (CBF)-(T6) | T6_12 months later
  Hemoencephalography (HEG) will be measure by Bioland, the unit is ratio A/B
6 minutes walk test-(T1) | T1-Baseline
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation.
6 minutes walk test-(T2) | T2-1 month later
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation.
6 minutes walk test-(T3) | T3-2 months later
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation.
6 minutes walk test-(T4) | T4-3 months later
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation.
6 minutes walk test-(T5) | T5-6 months later
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation.
6 minutes walk test-(T6) | T6-12 months later
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation.
Cardio force index (CFI)-(T1) | T1-Baseline
  CFI was measured by Bioharness device. The ratio is HR/peak activity. CFI is the index of cardiac force, correlated to VO2 max and can predict the physiological status of physical activity. The heart rate, respiratory rate, distance of walking/ exercise and angular acceleration are also be measured by Bioharness device in the same time to calculate the CFI.
Cardio force index (CFI)-(T2) | T2-1 month later
  CFI was measured by Bioharness device. The ratio is HR/peak activity. CFI is the index of cardiac force, correlated to VO2 max and can predict the physiological status of physical activity. The heart rate, respiratory rate, distance of walking/ exercise and angular acceleration are also be measured by Bioharness device in the same time to calculate the CFI.
Cardio force index (CFI)-(T3) | T3-2 month later
  CFI was measured by Bioharness device. The ratio is HR/peak activity. CFI is the index of cardiac force, correlated to VO2 max and can predict the physiological status of physical activity. The heart rate, respiratory rate, distance of walking/ exercise and angular acceleration are also be measured by Bioharness device in the same time to calculate the CFI.
Cardio force index (CFI)-(T4) | T4-3 months later
  CFI was measured by Bioharness device. The ratio is HR/peak activity. CFI is the index of cardiac force, correlated to VO2 max and can predict the physiological status of physical activity. The heart rate, respiratory rate, distance of walking/ exercise and angular acceleration are also be measured by Bioharness device in the same time to calculate the CFI.
Cardio force index (CFI)-(T5) | T5-6 months later
  CFI was measured by Bioharness device. The ratio is HR/peak activity. CFI is the index of cardiac force, correlated to VO2 max and can predict the physiological status of physical activity. The heart rate, respiratory rate, distance of walking/ exercise and angular acceleration are also be measured by Bioharness device in the same time to calculate the CFI.
Cardio force index (CFI)-(T6) | T6-12 months later
  CFI was measured by Bioharness device. The ratio is HR/peak activity. CFI is the index of cardiac force, correlated to VO2 max and can predict the physiological status of physical activity. The heart rate, respiratory rate, distance of walking/ exercise and angular acceleration are also be measured by Bioharness device in the same time to calculate the CFI.

SECONDARY OUTCOMES:
Cognitive function-(T1) | T1-Baseline
  Cognitive function will be measured by the Mini-Mental State Exam (MMSE )instrument. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function ... school (but not a graduate of), a score on the MMSE of 24 or below means cognitive impairment.
Cognitive function-(T2) | T2-1month later
  Cognitive function will be measured by the Mini-Mental State Exam (MMSE )instrument. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function ... school (but not a graduate of), a score on the MMSE of 24 or below means cognitive impairment.
Cognitive function-(T3) | T3-2month later
  Cognitive function will be measured by the Mini-Mental State Exam (MMSE )instrument. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function ... school (but not a graduate of), a score on the MMSE of 24 or below means cognitive impairment.
Cognitive function-(T4) | T4-3month later
  Cognitive function will be measured by the Mini-Mental State Exam (MMSE )instrument. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function ... school (but not a graduate of), a score on the MMSE of 24 or below means cognitive impairment.
Cognitive function-(T5) | T5-6months later
  Cognitive function will be measured by the Mini-Mental State Exam (MMSE )instrument. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function ... school (but not a graduate of), a score on the MMSE of 24 or below means cognitive impairment.
Cognitive function-(T6) | T6-12months later
  Cognitive function will be measured by the Mini-Mental State Exam (MMSE )instrument. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function ... school (but not a graduate of), a score on the MMSE of 24 or below means cognitive impairment.
Brain single photon emission computed tomography (SPECT)-(T1) | T1_Baseline
  brain Single Photon Emission Computed Tomography (SPECT) imaging has developed a substantial, evidence-based foundation and is now recommended by professional societies for numerous indications relevant to psychiatric practice.
Brain single photon emission computed tomography (SPECT)-(T4) | T4_6 months later
  brain Single Photon Emission Computed Tomography (SPECT) imaging has developed a substantial, evidence-based foundation and is now recommended by professional societies for numerous indications relevant to psychiatric practice.

OTHER OUTCOMES:
depression status-(T1) | T1-Baseline
  Depression will be measured by Beck depression index (BDI). The BDI scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. A score is assigned by totaling all items (after reversing the positive mood items]. The possible range for the 21-item scale is 0 to 63, and a cut off score of 16 or higher indicates the presence of significant depressive symptoms.
depression status-(T2) | T2-1 month later
  Depression will be measured by Beck depression index (BDI). The BDI scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. A score is assigned by totaling all items (after reversing the positive mood items]. The possible range for the 21-item scale is 0 to 63, and a cut off score of 16 or higher indicates the presence of significant depressive symptoms.
depression status-(T3) | T3-2 months later
  Depression will be measured by Beck depression index (BDI). The BDI scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. A score is assigned by totaling all items (after reversing the positive mood items]. The possible range for the 21-item scale is 0 to 63, and a cut off score of 16 or higher indicates the presence of significant depressive symptoms.
depression status-(T4) | T4-3 months later
  Depression will be measured by Beck depression index (BDI). The BDI scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. A score is assigned by totaling all items (after reversing the positive mood items]. The possible range for the 21-item scale is 0 to 63, and a cut off score of 16 or higher indicates the presence of significant depressive symptoms.
depression status-(T5) | T5-6 months later
  Depression will be measured by Beck depression index (BDI). The BDI scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. A score is assigned by totaling all items (after reversing the positive mood items]. The possible range for the 21-item scale is 0 to 63, and a cut off score of 16 or higher indicates the presence of significant depressive symptoms.
depression status-(T6) | T6-12 months later
  Depression will be measured by Beck depression index (BDI). The BDI scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. A score is assigned by totaling all items (after reversing the positive mood items]. The possible range for the 21-item scale is 0 to 63, and a cut off score of 16 or higher indicates the presence of significant depressive symptoms.
Quality of life-(T1): WHOQOL-BREF | T1-Baseline
  Quality of life will be measured by World Health organization quality of life (WHOQOL) instrument. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items.The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Quality of life-(T2): WHOQOL-BREF | T2-1 month later
  Quality of life will be measured by World Health organization quality of life (WHOQOL) instrument. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items.The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Quality of life-(T3): WHOQOL-BREF | T3-2 month later
  Quality of life will be measured by World Health organization quality of life (WHOQOL) instrument. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items.The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Quality of life-(T4): WHOQOL-BREF | T4-3 months later
  Quality of life will be measured by World Health organization quality of life (WHOQOL) instrument. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items.The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Quality of life-(T5): WHOQOL-BREF | T5- 6 months later
  Quality of life will be measured by World Health organization quality of life (WHOQOL) instrument. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items.The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Quality of life-(T6): WHOQOL-BREF | T6- 12 months later
  Quality of life will be measured by World Health organization quality of life (WHOQOL) instrument. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items.The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
resilience status-(T1) | T1-Baseline
  Resilience will be measured by Resilience scale for adult scale. The Resilience Scale for Adults (RSA) (Friborg et al., 2003) is a 37-item scale that measures resilience as healthy adaptation and personal competence during exposure to significant adversity, trauma, or stress.
resilience status-(T2) | T2-1 month later
  Resilience will be measured by Resilience scale for adult scale. The Resilience Scale for Adults (RSA) (Friborg et al., 2003) is a 37-item scale that measures resilience as healthy adaptation and personal competence during exposure to significant adversity, trauma, or stress.
resilience status-(T3) | T3-2 month later
  Resilience will be measured by Resilience scale for adult scale. The Resilience Scale for Adults (RSA) (Friborg et al., 2003) is a 37-item scale that measures resilience as healthy adaptation and personal competence during exposure to significant adversity, trauma, or stress.
resilience status-(T4) | T4-3 months later
  Resilience will be measured by Resilience scale for adult scale. The Resilience Scale for Adults (RSA) (Friborg et al., 2003) is a 37-item scale that measures resilience as healthy adaptation and personal competence during exposure to significant adversity, trauma, or stress.
resilience status-(T5) | T5-6 months later
  Resilience will be measured by Resilience scale for adult scale. The Resilience Scale for Adults (RSA) (Friborg et al., 2003) is a 37-item scale that measures resilience as healthy adaptation and personal competence during exposure to significant adversity, trauma, or stress.
resilience status-(T6) | T6-12 months later
  Resilience will be measured by Resilience scale for adult scale. The Resilience Scale for Adults (RSA) (Friborg et al., 2003) is a 37-item scale that measures resilience as healthy adaptation and personal competence during exposure to significant adversity, trauma, or stress.
Post-concussion symptom-(T1) | T1-Baseline
  post-concussion will be measured by the Rivermead post-concussion symptom scale.
Post-concussion symptom-(T2) | T2-1 month later
  post-concussion will be measured by the Rivermead post-concussion symptom scale.
Post-concussion symptom-(T3) | T3-2 months later
  post-concussion will be measured by the Rivermead post-concussion symptom scale.
Post-concussion symptom-(T4) | T4-3 months later
  post-concussion will be measured by the Rivermead post-concussion symptom scale.
Post-concussion symptom-(T5) | T5-6 months later
  post-concussion will be measured by the Rivermead post-concussion symptom scale.
Post-concussion symptom-(T6) | T6-12 months later
  post-concussion will be measured by the Rivermead post-concussion symptom scale.
Self-efficacy-(T1) | T1- Baseline
  Self-efficacy will be measured by the self-efficacy scale.
Self-efficacy-(T2) | T2- 1 month later
  Self-efficacy will be measured by the self-efficacy scale.
Self-efficacy-(T3) | T3- 2 months later
  Self-efficacy will be measured by the self-efficacy scale.
Self-efficacy-(T4) | T4- 3 months later
  Self-efficacy will be measured by the self-efficacy scale.
Self-efficacy-(T5) | T5- 6 months later
  Self-efficacy will be measured by the self-efficacy scale.
Self-efficacy-(T6) | T6- 12 months later
  Self-efficacy will be measured by the self-efficacy scale.
Sleep quality-(T1) | T1- Baseline
  Sleep quality will be measured by the Pittsburgh sleep quality scale and the Garmin vivosmart sleep records and its physiological recording.
Sleep quality-(T2) | T2- 1 month later
  Sleep quality will be measured by the Pittsburgh sleep quality scale and the Garmin vivosmart sleep records and its physiological recording.
Sleep quality-(T3) | T3- 2 months later
  Sleep quality will be measured by the Pittsburgh sleep quality scale and the Garmin vivosmart sleep records and its physiological recording.
Sleep quality-(T4) | T4- 3 months later
  Sleep quality will be measured by the Pittsburgh sleep quality scale and the Garmin vivosmart sleep records and its physiological recording.
Sleep quality-(T5) | T5- 6 months later
  Sleep quality will be measured by the Pittsburgh sleep quality scale and the Garmin vivosmart sleep records and its physiological recording.
Sleep quality-(T6) | T6- 12 months later
  Sleep quality will be measured by the Pittsburgh sleep quality scale and the Garmin vivosmart sleep records and its physiological recording.
Sport motivation Scale-(T1) | T1- baseline
  Sport motivation will be measure by the Sport Motivation Scale II (SMS-II)and exercise motivation interview. The 18-item SMS-II consists of six subscalesmeasuring amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Each subscale has three items. Participants were asked to respond to all the items on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true).
Sport motivation Scale-(T2) | T2- 1 month later
  Sport motivation will be measure by the Sport Motivation Scale II (SMS-II)and exercise motivation interview. The 18-item SMS-II consists of six subscalesmeasuring amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Each subscale has three items. Participants were asked to respond to all the items on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true).
Sport motivation Scale-(T3) | T3- 2 month later
  Sport motivation will be measure by the Sport Motivation Scale II (SMS-II)and exercise motivation interview. The 18-item SMS-II consists of six subscalesmeasuring amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Each subscale has three items. Participants were asked to respond to all the items on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true).
Sport motivation Scale-(T4) | T4- 3 month later
  Sport motivation will be measure by the Sport Motivation Scale II (SMS-II)and exercise motivation interview. The 18-item SMS-II consists of six subscalesmeasuring amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Each subscale has three items. Participants were asked to respond to all the items on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true).
Sport motivation Scale-(T5) | T5- 6 month later
  Sport motivation will be measure by the Sport Motivation Scale II (SMS-II)and exercise motivation interview. The 18-item SMS-II consists of six subscalesmeasuring amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Each subscale has three items. Participants were asked to respond to all the items on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true).
Sport motivation Scale-(T6) | T6- 12 month later
  Sport motivation will be measure by the Sport Motivation Scale II (SMS-II)and exercise motivation interview. The 18-item SMS-II consists of six subscalesmeasuring amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. Each subscale has three items. Participants were asked to respond to all the items on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true).

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsun Chiang, PhD, Principal Investigator — National Defense Medical Center
Locations (1):
- TSGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanderbeken I, Kerckhofs E. A systematic review of the effect of physical exercise on cognition in stroke and traumatic brain injury patients. NeuroRehabilitation. 2017;40(1):33-48. doi: 10.3233/NRE-161388. PMID 27814304
- [Background] Churchill JD, Galvez R, Colcombe S, Swain RA, Kramer AF, Greenough WT. Exercise, experience and the aging brain. Neurobiol Aging. 2002 Sep-Oct;23(5):941-55. doi: 10.1016/s0197-4580(02)00028-3. PMID 12392797
- [Background] Hassett LM, Moseley AM, Tate R, Harmer AR. Fitness training for cardiorespiratory conditioning after traumatic brain injury. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006123. doi: 10.1002/14651858.CD006123.pub2. PMID 18425937
- [Background] Snyder HR, Kaiser RH, Warren SL, Heller W. Obsessive-compulsive disorder is associated with broad impairments in executive function: A meta-analysis. Clin Psychol Sci. 2015 Mar;3(2):301-330. doi: 10.1177/2167702614534210. PMID 25755918
- [Background] Taylor JM, Montgomery MH, Gregory EJ, Berman NE. Exercise preconditioning improves traumatic brain injury outcomes. Brain Res. 2015 Oct 5;1622:414-29. doi: 10.1016/j.brainres.2015.07.009. Epub 2015 Jul 9. PMID 26165153
- [Background] Devine JM, Wong B, Gervino E, Pascual-Leone A, Alexander MP. Independent, Community-Based Aerobic Exercise Training for People With Moderate-to-Severe Traumatic Brain Injury. Arch Phys Med Rehabil. 2016 Aug;97(8):1392-7. doi: 10.1016/j.apmr.2016.04.015. Epub 2016 May 20. PMID 27216223
- [Derived] Chen HJ, Ma CY, Lin LF, Chang CC, Hueng DY, Chang YC, Chiang HH. Can symptom-severity phenotypes identify depression risk after mild traumatic brain injury? A cluster-based approach. BMC Psychiatry. 2025 Nov 4;25(1):1054. doi: 10.1186/s12888-025-07512-w. PMID 41188789